CLINICAL TRIAL: NCT04141514
Title: Effects of Short-term Therapeutic Fasting on Nausea and Vomiting Due to Chemotherapy
Acronym: CHEMO-FAST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2019/CHU/03
Record Dates: First submitted 2019-10-23; First posted 2019-10-28 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Nausea Post Chemotherapy; Vomiting
MeSH Terms: conditions — Vomiting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): therapeutic fasting
  Interventions: Other: therapeutic fasting
- control group (No Intervention): usual alimentation

INTERVENTIONS:
Other: therapeutic fasting — fasting limited to daily 250 kcal during 3 days (day before chemotherapy, the D day of the chemotherapy and the day after chemotherapy)
  Arms: intervention group

SUMMARY:
This study aims to estimate the effect of the practice of a short-term partial fasting compared to a usual alimentation on nausea and vomiting within 5 days after the start of a chemotherapy session on 2 successive chemotherapy courses (4 sessions of chemotherapy) in patients starting treatment with highly emetogenic chemotherapy (ABVD or AVD protocol).

DETAILED DESCRIPTION:
Patients in fasting arm will practice partial fasting during 3 days (D-1, D1 (D day of chemotherapy) and D2) following a food guide during 4 chemotherapy sessions. Patients in usual alimentation arm will continue to take food as usual practice.

In each arm, patients will be interviewed at each chemotherapy sessions about nausea and vomiting (number and intensity of nausea and vomiting, treatments taken). Denutrition, quality of life improvement, compliance to partial fasting, treatment response will be evaluate too.

ELIGIBILITY:
Inclusion Criteria:

* patient starting a treatment by chemotherapy ABVD or AVD
* patient affiliated to a social security scheme
* patient who gives his informed consent before any procedure related to the study

Exclusion Criteria:

* patient with diabetes
* patient with recent gastric ulcer
* patient with low BMI (less than 18,5 for patients under 70 or less than 21 for patient over 70)
* albuminemia <35
* patient wiht loss weight > 10% in 6 months
* pregnant or lactating women
* chronic alcoholism
* unable to understand the objectives and risks of the study
* patient with psychiatric desorder, under guardianship or under judicial protection
* patient who cannot read

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-01-20 (Actual); Primary Completion 2024-11-19 (Estimated); Study Completion 2025-06-19 (Estimated)

PRIMARY OUTCOMES:
nausea and vomiting evaluation and quantification | Day 1 (first day of the chemotherapy cycle),
  Anti-emetic tool from MASCC (Multinational Association of Supportive Care in Cancer)
nausea and vomiting evaluation and quantification | day 2 of the chemotherapy cycle
  Anti-emetic tool from MASCC (Multinational Association of Supportive Care in Cancer)
nausea and vomiting evaluation and quantification | day 3 of the chemotherapy cycle
  Anti-emetic tool from MASCC (Multinational Association of Supportive Care in Cancer)
nausea and vomiting evaluation and quantification | day 4 of the chemotherapy cycle
  Anti-emetic tool from MASCC (Multinational Association of Supportive Care in Cancer)
nausea and vomiting evaluation and quantification | day 5 of the chemotherapy cycle
  Anti-emetic tool from MASCC (Multinational Association of Supportive Care in Cancer)

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Elora MUSSARD, Principal Investigator — CHU de La Réunion
Locations (1):
- CHU de la Réunion, Saint-Pierre, France

IPD SHARING:
Plan to Share IPD: No